CLINICAL TRIAL: NCT01863433
Title: A Phase IV, Single-Centre, Open-label Study to Evaluate the Immunogenicity and Safety of the 2013/2014 Formulation of a bioCSL Split Virion, Inactivated Influenza Vaccine in Healthy Volunteers Aged 18-60 Years
Brief Title: A Study to Assess the Immunogenicity and Safety of a Trivalent Influenza Vaccine Containing the 2013/2014 Formulation of Enzira® Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSLCT-TIV-13-84; 2013-001420-19 (EudraCT Number)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trivalent Influenza Vaccine (Experimental): The study vaccine is a sterile, thiomersal-free suspension containing 45 mcg total haemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2013/2014 influenza season). The vaccine will be administered by intramuscular or deep subcutaneous injection.
  Interventions: Biological: Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine

SUMMARY:
This is a study to assess the immune (antibody) response and safety of a bioCSL split virion, inactivated influenza vaccine containing the 2013/2014 formulation of Enzira® vaccine in healthy adult volunteers aged between 18 and 60 years.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged between 18 and 60 years at the time of vaccination.
* Females of child-bearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen for the duration of the study. Females of child-bearing potential must return a negative urine pregnancy test result prior to vaccination with the vaccine.

Exclusion Criteria:

* Known hypersensitivity to a previous vaccination with influenza vaccine or allergy to eggs, ovalbumin, chicken protein, neomycin, polymyxin, or any components of the vaccine.
* Clinical signs of an active infection.
* A clinically significant medical condition.
* Vaccination with a seasonal or experimental influenza virus vaccine in the 6 months preceding study entry.
* Females who are pregnant or lactating.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: bioCSL Head of Clinical Operations, Study Director — Seqirus
Locations (1):
- Study Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open label, non-randomized with single group assignment in healthy volunteers aged 18 to 60 years.
Groups:
- Trivalent Influenza Vaccine: Healthy volunteers aged between 18 and 60 years received a single 0.5 mL dose of Trivalent Influenza Vaccine by intramuscular or subcutaneous injection.
Period: Overall Study
Arm/Group | Trivalent Influenza Vaccine
Started | 120
Completed | 119 (1 subject was withdrawn from the study due to evidence of substance abuse.)
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trivalent Influenza Vaccine
Number analyzed (Participants) | 120
Age, Customized [Mean (Standard Deviation); unit: years] | 31.8 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Evaluable Participants Achieving Seroconversion or Significant Increase in Antibody Titre.
Description: As per the criteria specified in the CPMP/BWP/214/96 Note for Guidance on Harmonisation of Requirements for Influenza Vaccines. For haemagglutination inhibition (HI), seroconversion (H1N1, H3N2, and B influenza virus strains) is defined as achieving a post-vaccination titre of ≥ 40 for those participants with a pre-vaccination HI titre of < 10. A significant increase (H1N1, H3N2, and B influenza virus strains) is defined as a four-fold or greater increase in HI titre for those participants with a pre-vaccination HI titre of ≥ 10.
Time Frame: Approximately 21 days after vaccination
Population: The Evaluable Population includes all participants who were vaccinated with Trivalent Influenza Vaccine, provided both pre- and post-vaccination antibody titre results, did not use a prohibited medication as per the protocol, and were not excluded from the analysis according to the elimination criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trivalent Influenza Vaccine
Number analyzed (Participants) | 119
percentage of participants
  H1N1 strain | 79 [70.6 to 85.9]
  H3N2 strain | 79 [70.6 to 85.9]
  B strain | 64.7 [55.4 to 73.2]

2. Primary Outcome: The Geometric Mean Fold Increase (GMFI) in Antibody Titre After Vaccination.
Description: GMFI (H1N1, H3N2, and B influenza virus strains) is defined as the geometric mean of the fold increases of post-vaccination antibody titre over the pre-vaccination antibody titre.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: fold increase
Arm/Group | Trivalent Influenza Vaccine
Number analyzed (Participants) | 119
fold increase
  H1N1 strain | 15.01 (4.27)
  H3N2 strain | 13.18 (4.494)
  B strain | 5.86 (3.461)

3. Primary Outcome: The Percentage of Evaluable Participants Achieving a HI Titre ≥ 40 or Single Radial Haemolysis (SRH) Area ≥ 25 mm2.
Description: For the H1N1, H3N2, and B influenza virus strains. Note: No SRH data were collected.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trivalent Influenza Vaccine
Number analyzed (Participants) | 119
percentage of participants
  H1N1 strain | 97.5 [92.8 to 99.5]
  H3N2 strain | 99.2 [95.4 to 100.0]
  B strain | 95.0 [89.3 to 98.1]

4. Secondary Outcome: Type and Frequency of Any Solicited Adverse Events (AEs)
Description: The percentage of participants reporting any solicited AEs.
Time Frame: During the 4 days after vaccination (Day 0 plus 3 days)
Population: The Safety Population included all participants who received Trivalent Influenza Vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Trivalent Influenza Vaccine
Number analyzed (Participants) | 120
percentage of participants
  Any solicited local AE | 52.5
  Induration > 50 mm | 0.8
  Erythema | 10
  Ecchymosis | 8.3
  Pain | 51.7
  Any solicited systemic AE | 19.2
  Temperature > 38°C for ≥ 24 hours | 0
  Chills | 10.8
  Malaise | 17.5

5. Secondary Outcome: Type and Frequency of Any Unsolicited AEs
Description: The percentage of participants reporting any unsolicited AEs. Unsolicited AEs included AEs other than those specifically solicited.
Time Frame: After vaccination until the end of the study; approximately 21 days.
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Trivalent Influenza Vaccine
Number analyzed (Participants) | 120
percentage of participants | 44.2

ADVERSE EVENTS:
Time Frame: For solicited AEs: During the 4 days after vaccination (Day 0 plus 3 days); For unsolicited AEs and serious AEs (SAEs): After vaccination until the end of the study (approximately 21 days).
Description: The other AEs presented include solicited and unsolicited AEs. The Safety Population included all participants who received Trivalent Influenza Vaccine and provided follow-up safety data.
Arm/Group | Trivalent Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 81/120
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trivalent Influenza Vaccine (N=120)
Chills (Gastrointestinal disorders) | 13 (13)
Injection site pain (General disorders) | 62 (64)
Malaise (General disorders) | 21 (21)
Injection site erythema (General disorders) | 12 (12)
Injection site haemorrhage (General disorders) | 10 (10)
Headache (Nervous system disorders) | 32 (41) — Unsolicited adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.